CLINICAL TRIAL: NCT02391012
Title: Fecal Transplantation for Inflammatory Bowel Disease
Acronym: FMT IBD
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: unable to recruit enough patients
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, NAFTALI TIMNA, MD, Meir Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0198-12-MMC
Record Dates: First submitted 2015-03-05; First posted 2015-03-18 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Inflammatory Bowel Disease
Keywords: Ulcerative colitis; Crohns disease; Microbial transplantation
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fecal microbial l transplantation (Experimental): patients with active colitis who will undergo treatment by fecal microbial transplantation
  Interventions: Biological: Fecal microbial l transplantation

INTERVENTIONS:
Biological: Fecal microbial l transplantation — infusion of preparation of fecal preparation from a healthy donor to a colitis patient
  Other Names: FMT

SUMMARY:
Fecal microbial treatment (FMT) is a treatment that utilizes the microbiota of a healthy intestine as a probiotic preparation. The feces of a healthy individual is fluidized and than inserted into the intestinal tract of a sick individual, assuming that the healthy flora will colonize and cure the intestine. There are reports of the efficacy of this treatment for inflammatory bowel disease but currently the numbers are small.

aim: To investigate whether use of FMT will bring improvement for colitis in IBD patients . Methods: The patients will undergo full colonoscopy, the stool preparation will be infused through the colonoscope during withdrawal of the instrument.

DETAILED DESCRIPTION:
Back ground: intestinal microbiota have a central role in disease pathogenesis, either in a form of a "permissive" role or as a direct pathogenic cause.

Clostridium difficile colitis; irritable bowel syndrome (IBS) and IBD have all been connected to a disturbance in the equilibrium of intestinal microbiome. But the causative mechanism is not yet known. (5-10) . Various bacteria including lactobacillus acidophilus and bifidobacterium bifidus are being empirically used as treatment for many intestinal ailments. The cause of inflammatory bowel disease in unknown but evidence is gathering that excessive immune reaction of intestinal immune system to microflora combined with a genetic predisposition are responsible for the chronic inflammation.

Fecal microbial treatment (FMT) is a treatment that utilizes the microbiota of a healthy intestine as a probiotic preparation. The feces of a healthy individual is fluidized and that inserted into the intestinal tract of a sick individual, assuming that the healthy flora will colonize and cure the intestine. Previous work had shown success in fecal transplantation as a treatment for clostridium difficile colitis. There are also reports of the efficacy of this treatment for inflammatory bowel disease but currently the numbers are small. A review by Anderson et al describes 17 studies reporting treatment of IBD by FMT. (12). In 9 cases it was done to treat IBD and in 8 cases for intestinal infection in IBD patients. Altogether 41 cases were reported , In some the FMT was inserted through a nasogastric tube directly to the duodenum, in some be colonoscopy and in some by an enema. A significant clinical improvement was reported in 19/25 patients. 13/17 stopped IBD treatment , 15/24 entered full clinical remission. In all 15 patients treated for infection the treatment was successful. No sever adverse effects were reported, Fever was developed in 8 cases and in one case there was exacerbation of colitis after treatment.

Primary aim: To investigate whether use of FMT will bring improvement of at least 2 points in partial mayo score in ulcerative colitis patients, or 70 points in CDAI of patients with Crohn's colitis. One month after FMT.

Improvement will be defined as:

For Ulcerative colitis: a decrease of at least 2 points in the partial mayo score, and a decrease of at least 1 point in endoscopic Mayo score.

For Crohn's disease: A decrease of at least 70 points in Crohn's disease activity index (CDAI) .

Materials and methods:

Study population: 40 patients aged 18-80 years, with histological and endoscopic diagnosis of ulcerative colitis or crohn's colitis who did not respond to either thiopurines or tumor necrosis factor (TNF) inhibitors.

Exacerbation will be defined as partial mayo score higher then 3, with either CRP higher than 0.5 or endoscopic mayo score >1 in ulcerative colitis and CDAI higher them 220 and C reactive protein (CRP) higher than 0.5 in Crohn's colitis.

Stool will be donated by the patients choice either from a relative, preferably a partner to minimize possible transference of an infective agent, alternatively samples will be ordered from "open biom".

Endoscopic disease activity will be defined as follows:

Endoscopic Mayo score:

* Normal or inactive disease: 0
* Mild disease (erythema, decreased vascular pattern, mild friability): 1
* Moderate disease (marked erythema, absent vascular pattern, friability, erosions): 2
* Severe disease (spontaneous bleeding, ulceration): 3

Simple endoscopic score Crohns disease (SES-CD):

Segments of intestine: Rectum,Sigmoid and left colon, Transverse colon,Right colon, Ileum for each segment the Presence of: ulcers,Ulcerated surface, Affected surface, Presence of narrowing, and number of affected segments will be evaluated and the total score sumed, The SES-CD will than be calculated as follows: TOTAL - 1.4 X (number of affected segments) = E-CDI

Inclusion criteria

Donor:

1. Signed informed consent
2. Basically healthy, no hospitalization in the last 6 months, no active malignant disease (with the exclusion of Basal cell skin tumor that was treated).
3. No antibiotic treatment in the last 6 months
4. Preferably a partner of the patient, or a relative leaving in the same house
5. No febrile illness in the last month
6. Normal laboratory tests including: blood count, liver and kidney function, negative hepatitis A immunoglobulin M (IgM), negative hepatitis C antibody, negative HbsAg, negative HIV , human T-lymphotropic virus (HTLV I/II), negative venereal disease research laboratory ( VDRL).
7. Stool tests: Negative stool culture, negative C. difficile toxins (A and B). Negative parasite microscopy. Fecal calprotectin.

Patient:

1. Signed informed consent
2. Inflammatory bowel disease diagnosed at least 3 months ago
3. Failure of either one immunomodulator of at least 3 months duration, or TNF inhibitor full induction treatment, or intolerance to either of these drugs.
4. Currently active disease, partial Mayo score ≥4 for ulcerative colitis (UC), or CDAI ≥200 for Crohn's disease (CD).
5. negative HIV , HTLV I/II, negative stool culture, Negative C diff toxin, negative cytomegalovirus ( CMV)

Treatment protocol:

1. Both donor and recipient will sign informed consent
2. Both donor and recipient will do the above mentioned laboratory tests, the investigator will verify that the results are negative.
3. Recipient will be prepared for colonoscopy with 3 liters of polyethylene glycol according to the routine protocol.
4. The donor will bring same day stool, alternatively, preparation from "open biom" will be used.
5. 200 gr stools will be mixed with sterile 200ml sodium chloride (NACL) 0.9% and then filtered to exclude large particles.
6. The patients will undergo full colonoscopy, the stool preparation will be infused through the colonoscope during withdrawal of the instrument.
7. If no improvement within 7 days, the patient will be offered the option of another FMT using enema prepared in a similar manner.
8. Patients will be instructed to maintain a high fiber diet,

Follow up:

On first colonoscopy:

Exact description of the length of the involved segment + Mayo visual score for UC and simple endoscopic score - CD (SES -CD) for Crohn's disease.

2 biopsies from each colonic segment: Rt colon, transverse colon, left colon, rectum.

Weekly partial Mayo score or Harvey Bradshow Index (HBI ) in the first month, then once a month for 6 months.

After 6 months repeat colonoscopy + biopsies + stool samples. Colonoscopy does not have to be complete but has to include the segment that was inflamed in the first colonoscopy.

At the time of colonoscopy blood tests including complete blood count (CBC), liver and kidney function, CRP, fecal calprotectin.

Microbiota profiles:

1. From both the donor and the recipient before FMT.
2. From the recipient: one month and 6 months after FMT. Stool samples will be frozen immediately at -20° and then transferred to the laboratory for microbiota analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Inflammatory bowel disease diagnosed at least 3 months ago
3. Failure of either one immunomodulator of at least 3 months duration, or TNF inhibitor full induction treatment, or intolerance to either of these drugs.
4. Currently active disease, partial Mayo score ≥4 for ulcerative colitis, or CDAI ≥200 for CD.
5. negative HIV , HTLV I/II, negative stool culture, Negative C diff toxin, negative CMV

Exclusion Criteria:

1. No informed consent
2. Non active inflammatory bowel disease.
3. Active infection in either the donor or the recipient,

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-04; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Improvement of disease activity index. | 4 weeks
  : a decrease of at least 2 points in the partial mayo score, and a decrease of at least 1 point in endoscopic Mayo score.
  For Crohn's disease: A decrease of at least 70 points in CDAI.

SECONDARY OUTCOMES:
improvement of endoscopic score | 4 weeks
  Improvement of at least one point in endoscopic score
Maintenance of remission/ improvement during follow up | 6 months
  Maintenance of remission/ improvement during follow up
Patients perspective of the treatment (do patients regard the treatment as acceptable) | 6 months
  do patients regard the treatment as acceptable
Cost estimation of the treatment | 6 months
  cost of treatment
side effects (presence of fever,or rise of 50% or more in the number of bowel movements) | 6 months
  monitoring side effects of treatment,specifically the presence of fever above 38ۨ c or a rise of 50% or more in the number of bowel movements during the first 3 days after the infusion

CONTACTS AND LOCATIONS:
Overall Officials: Timna Naftali, MD, Principal Investigator — Meir Medical Center
Locations (2):
- Israel (2):
  - Meir hospital, Kfar Saba
  - Gastroenterology institute Meir Hospital, Kfar Saba

REFERENCES:
- [Background] Anderson JL, Edney RJ, Whelan K. Systematic review: faecal microbiota transplantation in the management of inflammatory bowel disease. Aliment Pharmacol Ther. 2012 Sep;36(6):503-16. doi: 10.1111/j.1365-2036.2012.05220.x. Epub 2012 Jul 25. PMID 22827693